CLINICAL TRIAL: NCT06947798
Title: The Effect of Motivational Interviewing on Anthropometric Measurements, Eating Attitudes, and Cardiometabolic Index in Overweight and Obese Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Saltuklu Aile Sağlığı Merkezi (Other)
Responsible Party: Principal Investigator, ORHUN DÖNMEZ, Principal Investigator, Saltuklu Aile Sağlığı Merkezi
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Saltuklu ASM
Record Dates: First submitted 2025-04-17; First posted 2025-04-27 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Motivational Interviewing; Cardiometabolic Index; Obesity; Overweight (BMI > 25); Anthropometric Measurements; Eating Behavior Disorders
MeSH Terms: conditions — Obesity; Overweight | interventions — Motivational Interviewing; Diet; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Active Comparator): In addition to the procedures applied to the control group, the experimental group was also subjected to motivational interviewing
  Interventions: Behavioral: motivational interviewing; Other: Diet; Behavioral: Physical exercise
- Control (Active Comparator): The control group received a dietary intervention involving a daily caloric restriction and was instructed to engage in moderate-intensity aerobic exercise for 30 minutes, five times per week.
  Interventions: Other: Diet; Behavioral: Physical exercise

INTERVENTIONS:
Behavioral: motivational interviewing — motivational interviewing four times
  Arms: experimental group
Other: Diet — A calorie-restricted diet was implemented in both the intervention and control groups.
Behavioral: Physical exercise — A moderate-intensity aerobic exercise program, consisting of 30-minute sessions five days per week, was implemented in both groups

SUMMARY:
The Effect of Motivational Interviewing on Anthropometric Measurements, Eating Attitudes, and Cardiometabolic Index in Overweight and Obese Patients

DETAILED DESCRIPTION:
Participants were randomly assigned into two groups-an Intervention Group (n = 40) and a Control Group (n = 40)-using block randomization through the website "random.org." Data were collected using a Personal Information Form, the Eating Behavior Disorder Scale, Anthropometric Measurements (body weight, body mass index, waist circumference, waist/hip ratio), and the Cardiometabolic Index. Both groups received routine recommendations, which included a daily caloric restriction of 500 kcal and moderate-intensity aerobic exercise for 30 minutes, five days a week.Motivational interviewing was administered to the intervention group through individual sessions, held once every two weeks, for a total of four sessions, each lasting 15 minutes. The interviews were conducted in the Education Room of the Saltuklu Family Health Center. After the motivational interviewing intervention was completed, post-tests (Eating Behavior Disorder Scale, Anthropometric Measurements, and Cardiometabolic Index) were administered to both groups. All participants were followed for a period of three months.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) in the range of 25 to 34.9 kg/m² was considered as an inclusion criterion
* Being between 20 and 40 years of age (corresponding to the young adulthood period according to Erikson)

  -- Participants were required to be registered with the Saltuklu Family Health Center.
* Willingness to participate in the study and provision of informed consent were required

Exclusion Criteria:

* Current use of medications known to induce weight gain or loss
* Presence of a diagnosed chronic illness
* Pregnancy or being in the lactation period."

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
CMI | three months
  Cardiometabolic index

IPD SHARING:
Plan to Share IPD: Undecided